CLINICAL TRIAL: NCT02226159
Title: Surgery Prevention by Transforaminal Injection of Epidural Steroids for Cervical Radicular Pain (SPIES): a Randomized, Controlled Trial
Brief Title: Surgery Prevention by Transforaminal Injection of Epidural Steroids for Cervical Radicular Pain
Acronym: SPIES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Charlotte Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9086-14019
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Pain, Radiating
Keywords: cervical; radicular pain; transforaminal epidural steroid injections
MeSH Terms: conditions — Pain | interventions — Lidocaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Cervical transforaminal injection: 1.0 cc Lidocaine 1.0% with 1.0 cc normal saline
  Interventions: Drug: Lidocaine
- Lidocaine with Dexamethasone (Experimental): Cervical transforaminal injection: 1.0 cc Lidocaine 1.0% with 1.0 cc of Dexamethasone (10 mg/cc)
  Interventions: Drug: Lidocaine with Dexamethasone

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine
Drug: Lidocaine with Dexamethasone
  Other Names: Lidocaine; Dexamethasone
  Arms: Lidocaine with Dexamethasone

SUMMARY:
Cervical radicular pain is a common cause of disability and pain in the upper extremity and neck with an annual incidence of 83.2/100,000 (1). The initial treatment is conservative and includes relative rest, use of anti-inflammatory and analgesic medication, as well as physical therapy and home exercise. For patients who have persistent and significant symptoms, interventional pain management and surgical management are considered. Cervical epidural injections are the mainstay of the interventional, non-surgical modalities. They can be considered to provide short and long-term relief when disc herniation, foraminal stenosis or central canal stenosis pathology is identified. We are not aware of any published prospective, randomized, controlled, double-blinded studies demonstrating the efficacy of cervical transforaminal epidural steroid injections. However, the North American Spine Society (NASS) Review and Recommendation Statement states that based on the literature and expert opinion, a minimum of one or two cervical epidural steroid injections would be very appropriate in the treatment of a specific episode of cervical radicular pain.

The purpose of this study is to determine the effectiveness of cervical transforaminal epidural steroid injections in decreasing the need for an operation in patients with cervical radicular pain, otherwise considered to be operative candidates.

DETAILED DESCRIPTION:
Cervical radicular pain is a common cause of disability and pain in the upper extremity and neck with an annual incidence of 83.2/100,000 (1). The initial treatment is conservative and includes relative rest, use of anti-inflammatory and analgesic medication, as well as physical therapy and home exercise. For patients who have persistent and significant symptoms, interventional pain management and surgical management are considered. Cervical epidural injections are the mainstay of the interventional, non-surgical modalities. They can be considered to provide short and long-term relief when disc herniation, foraminal stenosis or central canal stenosis pathology is identified.

Cervical epidural injections can be performed by two different approaches, transforaminal and interlaminar. Transforaminal epidural injections allow delivery of medication to the ventral epidural space, while the interlaminar approach reaches the ventral epidural space in only 28% of injections (2-4). The results of cervical epidural injections remain controversial and their efficacy in decreasing the need for surgery in patients who would otherwise be operative candidates has not been thoroughly investigated. Studies have been limited by small sample sizes, lack of control groups, and lack of randomization. Kolstad et al reported that 23% (5/21) of patients waiting for cervical disc surgery cancelled surgery when assessed at four months after having a series of two cervical epidural injections (6). Lin et al reported that 63% (44/70) of patients who were deemed to be surgical candidates were able to avoid surgery with an average of 13-month follow up (7). Lee et al reported that over 80% of 98 patients evaluated with cervical radiculopathy were able to avoid surgery with a 2-year follow-up (8). Anderberg et al reported that there was no short-term difference in symptoms of cervical radiculopathy between patients who received transforaminal injections of steroid with local anesthetic versus saline with local anesthetic. However, this study did not evaluate whether the injections were successful in the patients avoiding surgery (11).

In terms of lumbar transforaminal epidural injections, Riew et al demonstrated that steroid injections obviated the need for surgery in patients with lumbar radiculopathy. Moreover, Reiw et al showed that steroid combined with local anesthetic was more effective than local anesthetic alone in a prospective, randomized, controlled, double-blinded study (9). Riew et al later studied the efficacy of cervical transforaminal epidural injections in the same fashion, but the findings were not statistically significant (p<0.35) and not published (10).

We are not aware of any published prospective, randomized, controlled, double-blinded studies demonstrating the efficacy of cervical transforaminal epidural steroid injections. However, the North American Spine Society (NASS) Review and Recommendation Statement states that based on the literature and expert opinion, a minimum of one or two cervical epidural steroid injections would be very appropriate in the treatment of a specific episode of cervical radicular pain. This literature also suggests that a maximum of four injections can be used within six months, assuming there was a positive response and improvement seen with the previous injections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have cervical radicular pain without significant neurologic deficit (neurologic deficit is defined as manual muscle testing less than 3/5), MRI/CT findings of neural compression (neural compression is defined as disc herniation or central or foraminal spinal stenosis),
* Failed 6 weeks of conservative treatment (conservative treatment is defined as relative rest, home exercise, physical therapy, and use of anti-inflammatory and/or analgesic medications),
* Deemed to be good operative candidates by spine surgeons (patients with MRI/CT findings of neural compression with concordant symptoms) and had agreed to possible operative intervention

Exclusion Criteria:

* History of

  1. acute trauma,
  2. diabetes (type I or type II),
  3. active infection
* Active progressive neurological deficit (neurologic is deficit defined as manual muscle testing less than 3/5),
* Medical condition that may affect the cervical spine neurological exam and/or pain assessment (e.g. peripheral neuropathy),
* Bilateral disease,
* More than one cervical level requiring injection,
* Bleeding disorders or other medical contraindications to the injection procedure,
* Absence of substantial radicular pain (radicular pain is defined as arm pain greater than neck pain),
* Involvement in workers' compensation claim, or any litigation related to neck injury.
* Patients who are pregnant, or who plan to become pregnant in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Bhagia, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Radhakrishnan K, Litchy WJ, O'Fallon WM, Kurland LT. Epidemiology of cervical radiculopathy. A population-based study from Rochester, Minnesota, 1976 through 1990. Brain. 1994 Apr;117 ( Pt 2):325-35. doi: 10.1093/brain/117.2.325. PMID 8186959
- [Background] Stojanovic MP, Vu TN, Caneris O, Slezak J, Cohen SP, Sang CN. The role of fluoroscopy in cervical epidural steroid injections: an analysis of contrast dispersal patterns. Spine (Phila Pa 1976). 2002 Mar 1;27(5):509-14. doi: 10.1097/00007632-200203010-00011. PMID 11880836
- [Background] Strub WM, Brown TA, Ying J, Hoffmann M, Ernst RJ, Bulas RV. Translaminar cervical epidural steroid injection: short-term results and factors influencing outcome. J Vasc Interv Radiol. 2007 Sep;18(9):1151-5. doi: 10.1016/j.jvir.2007.06.011. PMID 17804778
- [Background] Lieberman R, Dreyfuss P, Baker R. Fluoroscopically guided interlaminar cervical epidural injections. Arch Phys Med Rehabil. 2003 Oct;84(10):1568-9; author reply 1569. doi: 10.1016/j.apmr.2003.08.072. No abstract available. PMID 14594016
- [Background] Manchikanti L, Falco FJ, Diwan S, Hirsch JA, Smith HS. Cervical radicular pain: the role of interlaminar and transforaminal epidural injections. Curr Pain Headache Rep. 2014 Jan;18(1):389. doi: 10.1007/s11916-013-0389-9. PMID 24338702
- [Background] Kolstad F, Leivseth G, Nygaard OP. Transforaminal steroid injections in the treatment of cervical radiculopathy. A prospective outcome study. Acta Neurochir (Wien). 2005 Oct;147(10):1065-70; discussion 1070. doi: 10.1007/s00701-005-0542-2. Epub 2005 Jun 9. PMID 15924210
- [Background] Lin EL, Lieu V, Halevi L, Shamie AN, Wang JC. Cervical epidural steroid injections for symptomatic disc herniations. J Spinal Disord Tech. 2006 May;19(3):183-6. doi: 10.1097/01.bsd.0000190558.13248.e1. PMID 16770215
- [Background] Lee SH, Kim KT, Kim DH, Lee BJ, Son ES, Kwack YH. Clinical outcomes of cervical radiculopathy following epidural steroid injection: a prospective study with follow-up for more than 2 years. Spine (Phila Pa 1976). 2012 May 20;37(12):1041-7. doi: 10.1097/BRS.0b013e31823b4d1f. PMID 22024908
- [Background] Riew KD, Yin Y, Gilula L, Bridwell KH, Lenke LG, Lauryssen C, Goette K. The effect of nerve-root injections on the need for operative treatment of lumbar radicular pain. A prospective, randomized, controlled, double-blind study. J Bone Joint Surg Am. 2000 Nov;82(11):1589-93. doi: 10.2106/00004623-200011000-00012. PMID 11097449
- [Background] Anderberg L, Annertz M, Persson L, Brandt L, Saveland H. Transforaminal steroid injections for the treatment of cervical radiculopathy: a prospective and randomised study. Eur Spine J. 2007 Mar;16(3):321-8. doi: 10.1007/s00586-006-0142-8. Epub 2006 Jul 12. PMID 16835737

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine: Cervical transforaminal injection: 1.0 cc Lidocaine 1.0% with 1.0 cc normal saline
  Lidocaine
- Lidocaine With Dexamethasone: Cervical transforaminal injection: 1.0 cc Lidocaine 1.0% with 1.0 cc of Dexamethasone (10 mg/cc)
  Lidocaine with Dexamethasone
Period: Overall Study
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Started | 33 | 32
Completed | 27 | 26
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Lidocaine With Dexamethasone | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [44 to 58] | 53.5 [46 to 62] | 52 [45 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 24 | 50
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 16 | 22 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53
Verbal Numeric Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — On a scale of 1-10 with 10 indicating the greatest among of pain
  units on a scale | 5 [5 to 7] | 7 [5 to 8] | 6.5 [5 to 8]
Neck Disability Index [Median (Inter-Quartile Range); unit: units on a scale] — Scored from 0-50, with 50 indicating the greatest amount of disability
  units on a scale | 33 [26 to 40] | 35 [24 to 48] | 34 [26 to 44]
Patient Satisfaction [Median (Inter-Quartile Range); unit: units on a scale] — Scored from 0-10 with 10 indicating the greatest among of patient satisfaction
  units on a scale | 5 [3 to 5] | 3 [2 to 5] | 3.5 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Avoidance of Neck Surgery
Description: The primary outcome variable is the avoidance of surgery. Treatment success is defined as the avoidance of surgery, while treatment failure is defined as having surgery due to failure of the injection treatment to alleviate pain and improve function over the 12 months they are being followed for purposes of this study. Avoided neck surgery noted as 'Yes'; avoided neck surgery 'No' the patient had neck surgery.
Time Frame: 12 months after the first injection
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
Participants
  No(had surgery) | 24 | 20
  Yes (Did not have surgery) | 3 | 6

2. Secondary Outcome: Disability
Description: Neck Disability Index (NDI) - The NDI consists of 10 questions. Each of the 10 items is scored from 0 (minimum) - 5(maximum). The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score (i.e. a score of 50 indicates 100% disability). Scores are reported as the percentage (i.e. 100 is the max score for data presented).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
units on a scale | 25.2 (14.1) | 22.8 (17.2)

3. Secondary Outcome: Numeric Pain Scre
Description: Verbal Numeric Pain Scale (VNPS) -Scaled 0-10 with 10 being worst imaginable pain and 0 being no pain
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 3.7 (2.8) | 3.8 (2.9)

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with the treatment. Scale is an inverse of verbal numeric pain score. A 0 on VNPS equates to a 10 on patient satisfaction, 10 on VNPS equates to 0 on patient satisfaction
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 6.3 (2.8) | 6.2 (2.9)

5. Secondary Outcome: Disability
Description: Neck Disability Index- The NDI consists of 10 questions. Each of the 10 items is scored from 0 (minimum) - 5(maximum). The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score (i.e. a score of 50 indicates 100% disability). Scores are reported as the percentage (i.e. 100 is the max score for data presented).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
units on a scale | 25.1 (15.3) | 18.3 (18.4)

6. Secondary Outcome: Disability
Description: as for outcome 5
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
units on a scale | 19.4 (14.0) | 16.3 (17.5)

7. Secondary Outcome: Disability
Description: as for outcome 5
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
units on a scale | 16.4 (14.4) | 15.4 (10.2)

8. Secondary Outcome: Numeric Pain Score
Description: Verbal Numeric Pain Scale-Scaled 0-10 with 10 being worst imaginable pain and 0 being no pain
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 3.6 (2.4) | 3.4 (3.0)

9. Secondary Outcome: Numeric Pain Score
Description: Verbal Numeric Pain Scale-Scaled 0-10 with 10 being worst imaginable pain and 0 being no pain
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 3.0 (2.4) | 2.2 (2.8)

10. Secondary Outcome: Numeric Pain Score
Description: Verbal Numeric Pain Scale-Scaled 0-10 with 10 being worst imaginable pain and 0 being no pain
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 2.9 (2.8) | 3.2 (3.1)

11. Secondary Outcome: Patient Satisfaction
Description: as for outcome 4
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 6.4 (2.4) | 6.6 (3.0)

12. Secondary Outcome: Patient Satisfaction
Description: as for outcome 4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 7.0 (2.4) | 7.8 (2.8)

13. Secondary Outcome: Patient Satisfaction
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
Number analyzed (Participants) | 27 | 26
score on a scale | 7.2 (2.8) | 6.8 (3.1)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected at weeks 1, 2, 3, 4, and 12, then at 6 months and 12 months
Arm/Group | Lidocaine | Lidocaine With Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 3/27 | 9/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=27) | Lidocaine With Dexamethasone (N=26)
Numbness and tingling (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 3 (3)
Increased arm/neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
chest pain (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 2 (2)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hot/flushed feeling (General disorders) | 0 (0) | 1 (1)
Pain at injection site (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02226159/Prot_SAP_000.pdf